CLINICAL TRIAL: NCT03353285
Title: Effect of Follicle Flushing on Oocyte Fertilization Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Other Study IDs: number of flushes
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I: Group I= egg retrieved in the follicular fluid of the first aspirate (no flushing)
  Interventions: Procedure: intracytoplasmic sperm injection (ICSI)
- Group II: Group II= egg retrieved in the 1st-2nd flush
  Interventions: Procedure: intracytoplasmic sperm injection (ICSI)
- Group III: Group III= egg retrieved in the 3rd-5th flush
  Interventions: Procedure: intracytoplasmic sperm injection (ICSI)

INTERVENTIONS:
Procedure: intracytoplasmic sperm injection (ICSI) — All eggs will be fertilized by ICSI

SUMMARY:
The purpose of this study is to investigate the impact of follicular flushing on fertilization rate in women undergoing IVF treatment

DETAILED DESCRIPTION:
This will be a prospective observational study on the effect of follicular flushing on fertilization rate in women undergoing IVF treatment.

Oocytes from each woman will be allocated to one of three groups, depending on the aspirate or flush they are recovered from:

Group I= egg retrieved in the follicular fluid of the first aspirate (no flushing) Group II= egg retrieved in the 1st-2nd flush Group III= egg retrieved in the 3rd-5th flush

development and utilization. Pregnancy rates will be reported as a surrogate outcome.

ELIGIBILITY:
Inclusion Criteria:

* Up to 40 years old
* Both ovaries present
* Triggering final oocyte maturation using hCG or GnRH agonist

Exclusion Criteria:

* Egg donation
* PGD cases

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Women undergoing IVF treatment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | Day 1 post oocyte retrieval
  Number of fertilized eggs per oocyte retrieved

SECONDARY OUTCOMES:
Maturation rate | Day of oocyte retrieval
  Number of mature (MII) eggs per oocyte retrieved
Good quality embryos | Day 2 post oocyte retrieval
  Number of good quality embryos on Day 2
Blastocyst formation rate | Day 5 post oocyte retrieval
  Number of blastocysts on Day 5 per fertilized egg

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon G Lainas, Phd, Study Director — Eugonia
Locations (1):
- Eugonia, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] von Horn K, Depenbusch M, Schultze-Mosgau A, Griesinger G. Randomized, open trial comparing a modified double-lumen needle follicular flushing system with a single-lumen aspiration needle in IVF patients with poor ovarian response. Hum Reprod. 2017 Apr 1;32(4):832-835. doi: 10.1093/humrep/dex019. PMID 28333185
- [Background] Franasiak JM. Follicular flushing: time to look elsewhere to improve in vitro fertilisation outcomes? BJOG. 2017 Jul;124(8):1197. doi: 10.1111/1471-0528.14628. No abstract available. PMID 28276189
- [Background] Roque M, Sampaio M, Geber S. Follicular flushing during oocyte retrieval: a systematic review and meta-analysis. J Assist Reprod Genet. 2012 Nov;29(11):1249-54. doi: 10.1007/s10815-012-9869-9. Epub 2012 Oct 13. PMID 23065177